CLINICAL TRIAL: NCT03052556
Title: Prevalence and Persistence of Human Papillomavirus (HPV) and of Cervical Dysplasia in a Cohort of Women With Cystic Fibrosis
Brief Title: Human Papillomavirus and Cervical Dysplasia in Women With Cystic Fibrosis
Acronym: MUCOHPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL16_0703
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: cystic Fibrosis; cervical cancer; screening; human papilloma virus (HPV); pap smear test
MeSH Terms: conditions — Cystic Fibrosis; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort of women with cystic fibrosis (Other): Includable patients are adult women, transplanted or not, followed at Lyon CRCM (Centre de Ressources et de Compétences de la Mucoviscidose).
  Interventions: Procedure: Pap smear test and HPV test

INTERVENTIONS:
Procedure: Pap smear test and HPV test — Included women will attend a consultation with a gynaecologist. Pap smear test with HPV test will be performed. Samples collected by cervical scrape with a brush, will be prepared for liquid-based cytology. A sample of the sample will be used for research on HPV (Multiplex DNA PCR).
  This method allows detection of 35 different HPV genotypes: high risk (HPV-16, -18, -26, -31, -33, -35, -39, -45, -51, -52, 53, -56, -58, -59, -66, -68, -70, -73, -82, and -85); and low risk (HPV-6, -11, -40, -42, -43, -44, -54, -61, -62, -71, -72, -81, -83, -84, and -89).
  Patients with an initial abnormal pap smear or a positive HPV test will be monitored:
  * In case of an abnormal smear and / or positive HPV test, pap smear and HPV testing will be renewed every 6 months during the study period
  * In case of an abnormal smear:
  ASC-US: the attitude will depend on the result of the HPV test ASC-H, LSIL, HSIL, AGUS, AGC, AIS, carcinoma: a colposcopy will be performed

SUMMARY:
Background The main risk factor for cervical cancer is the infection by human papillomavirus (HPV), with several intermediate steps between HPV infection and cervical cancer. Cervical screening with pap smear test and HPV vaccination are effective preventions. A high frequency of HPV carriage and of cervical dysplasia have been described in transplanted women.

The majority of women with cystic fibrosis reach adulthood and some will face transplantation. Particular attention should therefore be paid to cervical screening. However, low adherence to screening recommendations was noted. In addition, preliminary data has found a high frequency of abnormal smears and of inflammatory aspect of the cervix in women with cystic fibrosis.

Objectives of the study The main objective of the study is to determine the prevalence of HPV carriage in a cohort of women with cystic fibrosis

The secondary objectives are:

* To study the factors associated with the prevalence of HPV (transplantation, smoking, age at first intercourse, number of sexual partners in the year, contraception, gravidity and parity, HPV vaccination)
* To describe and to compare with data in the general population, in hospital-based population, (and with data in transplanted population for transplanted women)

  1. the prevalence of HPV (and of different genotypes) infection, of cervical dysplasia, of vulvar/vaginal/cervical condylomatosis
  2. the rate of HPV persistence (> 12 months), the mean time of HPV clearance; rates of spontaneous regression / persistence / worsening of cervical dysplasia

Study design:

The study will last 24 months. Includable patients are adult women, transplanted or not, followed at Lyon CRCM. Included women will attend a consultation with a gynaecologist. Pap smear test (liquid phase cytology) and genomic DNA microarray assay enabling the detection of 35 different HPV genotypes will be performed.

Patients with an initial abnormal pap smear or a positive HPV test will be monitored:

* In case of an abnormal smear and / or positive HPV test, pap smear and HPV testing will be renewed every 6 months during the study period
* In case of an abnormal smear:

Atypical squamous cells of undetermined significance (ASC-US) : the attitude will depend on the result of the HPV test Atypical squamous cells - cannot exclude HSI L (ASC-H), Low-grade squamous intraepithelial lesion (LSIL), High-grade squamous intraepithelial lesion (HSIL), Atypical glandular cell of undetermined significance (AGUS) , Atypical glandular cells (AGC) , Adenoma carcinoma in situ (AIS), carcinoma: a colposcopy will be systematically performed

Expected results This study will help to determine the frequency of HPV infection and the pathogenic power of HPV in non-transplanted and in transplanted women with cystic fibrosis This data will help to sensitize health professionals on the importance of gynecological care and regular cervical screening, and on the importance of HPV vaccination.

In case of a high frequency of genital diseases linked to HPV, recommendations on gynecological monitoring procedures for women with cystic fibrosis could evolve.

ELIGIBILITY:
Inclusion Criteria:

* Female with Cystic fibrosis
* Age 18 years or older
* transplanted or non-transplanted
* Accepting the principle of a gynecological consultation and the principle of follow-up every 6 months in case of abnormal smear or positive HPV test
* Patient covered by health insurance

Exclusion Criteria:

* Age under 18
* Refusal to participate in the study
* Patient under tutorship / curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of HPV carriage | day 0
  Genomic DNA microarray assay enabling the detection of 35 different HPV genotypes will be performed.

SECONDARY OUTCOMES:
Rate of HPV persistence (> 12 months) | 12 months
  In case of a HPV positive test at inclusion, HPV tests will be repeated every 6 months during the study.
mean time of HPV clearance | 6 months, 12months, 18months and 24months
  In case of a HPV positive test at inclusion, HPV tests will be repeated every 6 months during the study.
Presence of factors associated with the prevalence of HPV | day 0
  factors studied are : transplantation, smoking, age at first intercourse, number of sexual partners in the year, contraception, gravidity and parity, HPV vaccination
Prevalence of cervical dysplasia or vulvar/vaginal/cervical condylomatosis | day 0
  Gynecological clinical examination with pap smear test will be performed at inclusion. The Bethesda system will be used for reporting Pap smear results. In case of abnormal pap smear, a colposcopy will be performed, with biopsies if indicated.
Rate of spontaneous regression of cervical dysplasia | 12 months and 24 months
  In case of high cervical dysplasia, usual recommended management will be executed. In case of low grade dysplasia (with concordant pap smear test and satisfactory colposcopy), a follow-up by colposcopy/biopsy will be performed every 6 months during the study
Rate of persistence of cervical dysplasia | 12 months and 24 months
  In case of high cervical dysplasia, usual recommended management will be executed. In case of low grade dysplasia (with concordant pap smear test and satisfactory colposcopy), a follow-up by colposcopy/biopsy will be performed every 6 months during the study
Rate of worsening of cervical dysplasia | 12 months and 24 months
  In case of high cervical dysplasia, usual recommended management will be executed. In case of low grade dysplasia (with concordant pap smear test and satisfactory colposcopy), a follow-up by colposcopy/biopsy will be performed every 6 months during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie oncologique - Centre Hospitalier Lyon Sud, Pierre-Bénite, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rousset-Jablonski C, Mekki Y, Denis A, Reynaud Q, Nove-Josserand R, Durupt S, Touzet S, Perceval M, Ray-Coquard I, Golfier F, Durieu I. Human papillomavirus prevalence, persistence and cervical dysplasia in females with cystic fibrosis. J Cyst Fibros. 2023 May;22(3):505-514. doi: 10.1016/j.jcf.2022.11.005. Epub 2022 Dec 14. PMID 36526553